CLINICAL TRIAL: NCT05595850
Title: A Mindful Community for People With ALS and Their Primary Caregivers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Harvard University (Other)
Collaborators: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Ellen Langer, Principal Investigator, Harvard University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB20-0629
Record Dates: First submitted 2022-09-12; First posted 2022-10-27 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Amyotrophic Lateral Sclerosis; Caregiver Burden
Keywords: Mindfulness; Quality of Life
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Caregiver Burden | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness (Experimental): Three-week online mindfulness course followed by one-month social community online interaction.
  Interventions: Behavioral: Mindfulness
- Mindful Learning (Active Comparator): Three-week online mindful learning course followed by one-month social community online interaction
  Interventions: Behavioral: Mindful Learning

INTERVENTIONS:
Behavioral: Mindfulness — Online non-meditation mindfulness program
  Arms: Mindfulness
Behavioral: Mindful Learning — Online learning program
  Arms: Mindful Learning

SUMMARY:
The psychological impact of ALS on patients and caregivers is high, significantly affecting their quality of life (QOL). Despite this impact, there is not much research about psychological interventions that could reduce psychological distress and improve QOL.

The efficacy of mindfulness-based treatments for the improvement of QOL was previously demonstrated by the investigator's group. Despite preliminary positive results, treatment efficacy tends to weaken over time. The investigators believe that a robust solution to maintain efficacy is to maximize the utilization of technology and emerging social platforms, establishing a "mindful community" to promote and continuously reinforce mindfulness.

This project's primary aims are 1) to develop a "mindful" online community of people with ALS and their caregivers, and 2) to test its efficacy in QOL improvement. This two-part intervention consists of 1) optimizing the investigator's prior e-learning platform with a three-week program including cognitive exercises, videos and lectures to increase participants' mindfulness; and 2) involving participants in a "mindfulness community" within a social sharing forum. Assessments will be performed before and immediately post-treatment as well as 3- and 6-months post-program comparing subjects undergoing the intervention to a control group.

ELIGIBILITY:
Inclusion Criteria:

For the ALS patients

* a definite, probable, laboratory-supported, or possible ALS by revised El-Escorial criteria
* they must have the physical ability, with or without adaptive devices, to use a smartphone, a tablet, or a computer
* have access to the Internet.

For the caregivers

* be the person who resides with the ALS patient and is the major provider of unpaid care and assistance (typically, the spouse or another close relative)
* s/he must be able to use the application
* have access to the Internet.

Exclusion criteria

- Using shared devices. Patients and caregivers should have their own devices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-10-12 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
ALS Specific QOL Short Form Quality of Life (ALSSQOL-SF) - For PALS (Persons with ALS) | 3 months
  The ALSSQOL-SF is a 20 item quality of life instrument for patients. It has a 0-10 rating scale with higher scores denoting higher QOL.
World Health Organization Quality of Life (Brief) WHO-QoL BREF - For Caregivers of PALS | 3 months
  The WHO-QoL BREF is a 26 item quality of life scale covering four domains of QOL. Each item is scored from 1-5 with higher response employing a higher quality of life. Items are scored from 1-5

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | 3 weeks, 3 months, 6 months after joining
  The HADS measures anxiety and depression in a general medical population of patients. It has seven items each for depression and anxiety sub scales. Scoring ranges from 0 to 3, with 3 denoting the highest anxiety or depression level. A total sub scale score of over 8 out of 21 denotes considerable symptoms of either.
Functional Status | 3 weeks, 3 months, 6 months after joining
  Self-Administered Functional Rating Scale Revised
Zarit Burden Interview | 3 weeks, 3 months, 6 months after joining
  The ZBI consists of 22 items rated on a 5-point Likert scale that ranges from 0 (never) to 4 (nearly always) with the sum of scores ranging between 0-88. Higher scores indicate greater burden. A score of 17 or more has been considered high burden.
ALS Specific QOL Short Form Quality of Life (ALSSQOL-SF) | 3 weeks, 3 months, 6 months after joining
  The ALSSQOL-SF is a 20 item quality of life instrument for patients. It has a 0-10 rating scale with higher scores denoting higher QOL.
World Health Organization Quality of Life (Brief) WHO-QoL BREF | 3 weeks, 3 months, 6 months after joining
  The WHO-QoL BREF is a 16 item quality of life scale covering four domains of QOL. Each item is scored from 1-5 with higher response employing a higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Langer, PhD, Principal Investigator — Harvard U
Locations (1):
- Harvard University, Cambridge, Massachusetts, United States